CLINICAL TRIAL: NCT04713254
Title: Interventional, Open-label, One-sequence Study to Investigate the Effects of Lu AG06466 on the Pharmacokinetics of the Cytochrome P450 Substrates Midazolam (CYP3A4), Bupropion (CYP2B6), and Metoprolol (CYP2D6) in Healthy Young Men and Women
Brief Title: Drug Drug Interaction Study With Lu AG06466 in Young Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19353A
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Metoprolol; Bupropion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lu AG06466 (Experimental)
  Interventions: Drug: Lu AG06466; Other: Midazolam; Other: Metoprolol; Other: Bupropion

INTERVENTIONS:
Drug: Lu AG06466 — 10, 20, 30 mg/day oral capsules on Day 5-18
Other: Midazolam — 4 mg syrup, oral single dose on Day 1 and Day 15
Other: Metoprolol — 100 mg tablets, oral single dose on Day 1 and Day 15
Other: Bupropion — 100 mg tablets, oral single dose on Day 3 and Day 17

SUMMARY:
The purpose of this study is to evaluate the effect of repeated doses of the drug Lu AG06466 on the exposure of metoprolol, midazolam and bupropion

DETAILED DESCRIPTION:
On Day 1, midazolam and metoprolol will be dosed as an oral single-dose cocktail and PK sampling will be performed for 48 hours.

On Day 3, bupropion will be dosed as a single oral dose and PK sampling will be performed for 48 hours.

On Days 5-18, subjects will be dosed with Lu AG06466 once daily.

On Day 15, midazolam and metoprolol will be dosed as an oral single-dose cocktail and PK sampling will be performed for 48 hours.

On Day 17, bupropion will be dosed as a single oral dose and PK sampling will be performed for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.5 to 30 kg/m2 (inclusive) at the Screening and Baseline Visits

Exclusion Criteria:

* The subject has any concurrent disorder that may affect the pharmacological target or absorption, distribution, or elimination of the investigational medicinal product.

Other in- and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
AUC 0-inf for midazolam | Day 1 and Day 15
  Area under the midazolam plasma concentration-time curve from zero to infinity
AUC 0-inf for metoprolol | Day 1 and Day 15
  Area under the metoprolol plasma concentration-time curve from zero to infinity
AUC 0-inf for bupropion | Day 3 and Day 17
  Area under the bupropion plasma concentration-time curve from zero to infinity
Cmax for midazolam | Day 1 and Day 15
  Maximum observed plasma concentration for midazolam
Cmax for metoprolol | Day 1 and Day 15
  Maximum observed plasma concentration for metoprolol
Cmax for bupropion | Day 3 and Day 17
  Maximum observed plasma concentration for bupropion

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance Dallas CRU, Dallas, Texas, United States